CLINICAL TRIAL: NCT06900036
Title: Radiographic Evaluation in Alveolar Preservation Using Platelet-rich Fibrin. Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Cuenca (Other)
Responsible Party: Principal Investigator, ROCIO MAGDALENA MOLINA BARAHONA, Oral and Maxillofacial Radiologist, Universidad Católica de Cuenca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEISH - UCACUE - 031
Record Dates: First submitted 2025-03-15; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Alveolar Bone Resorption; Preserving the Alveolar Ridge
Keywords: Bone Regeneration; Tooth Socket; oral surgery; Platelet-rich fibrin; CBCT
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet-Rich Fibrin (PRF) Application for Alveolar Preservation (Experimental): This arm involves the application of Platelet-Rich Fibrin (PRF) immediately after premolar extraction to evaluate its effectiveness in preserving alveolar bone structure and enhancing bone regeneration. PRF is a natural, autologous biomaterial obtained from the patient's own blood, promoting wound healing, bone preservation, and tissue regeneration.
  Interventions: Procedure: Platelet-Rich Fibrin (PRF) Application for Alveolar Preservation
- Control Group - Natural Healing (No PRF Application) (No Intervention): This arm represents the control group, where participants undergo standard premolar extraction without the application of platelet-rich fibrin (PRF). This allows for a direct comparison to assess the effectiveness of PRF in preserving alveolar bone and enhancing healing.

INTERVENTIONS:
Procedure: Platelet-Rich Fibrin (PRF) Application for Alveolar Preservation — This intervention involves the application of platelet-rich fibrin (PRF) in the extraction socket following premolar extraction to assess its effectiveness in alveolar bone preservation. PRF is a biological autologous material derived from the patient's own blood, promoting bone regeneration, wound healing, and tissue repair.
  Arms: Platelet-Rich Fibrin (PRF) Application for Alveolar Preservation

SUMMARY:
This randomized controlled trial is designed to assess the use of platelet-rich fibrin (PRF), a biomaterial derived from a participant's own blood, in alveolar ridge preservation following premolar extraction for orthodontic purposes. Participants aged 17 to 38 years requiring premolar extractions will be randomly assigned to receive either PRF application or natural healing without intervention. Cone beam computed tomography (CBCT) will be used to evaluate changes in alveolar bone dimensions and density at 30 and 120 days post-extraction. Measurements will be taken at standardized vertical levels (1 mm, 3 mm, and 5 mm apical to the crest) to analyze bone height, width, and density over time.

DETAILED DESCRIPTION:
This study is a randomized controlled clinical trial designed to investigate the application of platelet-rich fibrin (PRF) in post-extraction sites following orthodontically indicated premolar removals. PRF is prepared from autologous blood and applied to extraction sockets in the experimental group, while the control group undergoes standard physiological healing. Cone beam computed tomography (CBCT) will be used to obtain quantitative data on alveolar bone structure at baseline, 30 days, and 120 days post-extraction. The study will assess changes in bone height, horizontal ridge width at defined depths, and bone tissue density using standardized imaging protocols. This design allows for objective comparison between treated and untreated sites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with no systemic diseases.
* Age range: 17 to 38 years old.
* Orthodontic indication for premolar extraction (two maxillary or two mandibular premolars).
* Candidates for orthognathic surgery or extraction of impacted/retained teeth (e.g., third molars with a relationship to critical anatomical structures).
* Clinical justification for CBCT imaging instead of standard radiographic -techniques.

Exclusion Criteria:

* Patients with systemic diseases that may alter periodontal therapy outcomes.
* Platelet count below 200,000 mm³.
* Immunosuppressed patients.
* Pregnant or lactating women.
* Smokers.
* Patients taking medications that interfere with healing (e.g., bisphosphonates, corticosteroids, anticoagulants).

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Change in alveolar bone height (mm) at 30 and 120 days post-extraction as measured by CBCT | Baseline (immediately post-extraction), 30 days, and 120 days post-extraction.
  Alveolar bone height will be measured from the most apical point of the socket to the crestal margin using CBCT (cone beam computed tomography) scans at baseline (day of extraction), 30 days, and 120 days post-extraction. Measurements will be recorded in millimeters and compared between PRF-treated sites and control sites (no PRF). The mean difference in height over time will be calculated within and between groups.

SECONDARY OUTCOMES:
Change in alveolar bone depth (mm) at 1 mm, 3 mm, and 5 mm from crest, at 30 and 120 days post-extraction | Baseline, 30 days, and 120 days post-extraction.
  Bone depth (horizontal ridge width) will be assessed at three standardized vertical levels (1 mm, 3 mm, and 5 mm from the crestal margin) using CBCT imaging. Measurements will be performed bucco-lingually. Data will be reported as mean ± SD per time point and compared between PRF and control groups.
Bone tissue density (HU) at 30 and 120 days post-extraction measured via CBCT | Baseline, 30 days, and 120 days post-extraction.
  Bone density will be measured using Hounsfield Units (HU) within the center of the extraction socket. CBCT scans will be analyzed using imaging software calibrated for HU estimation. The average HU values will be compared between PRF-treated and control sockets to assess mineralization and bone quality.

CONTACTS AND LOCATIONS:
Overall Officials: ROCIO MAGDALENA MOLINA BARAHONA, Doctor of Dental Surgery (DDS), Principal Investigator — Universidad Católica de Cuenca; RENATA A AVECILLAS RODAS, Doctor of Dental Surgery (DDS), Study Chair — Universidad Católica de Cuenca
Locations (1):
- Universidad Catolica de Cuenca, Cuenca, Azuay, Ecuador

IPD SHARING:
Plan to Share IPD: Yes
Radiographic CBCT images (de-identified) Clinical measurements (bone height, depth, and quality) Demographic information (age, sex, general health status) Outcome measures (PRF effectiveness in alveolar preservation)
  Access Criteria:
  Available to qualified researchers upon request Requires a formal data access request and institutional agreement Compliance with ethical and privacy regulations
  Time Frame:
  Available upon study publication Accessible for at least five years post-publication
  Storage:
  Data will be stored in a secure university repository and potentially in public research databases.
  This plan ensures transparency, collaboration, and compliance with ICMJE guidelines for clinical research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start Date: Upon publication of study results End Date: At least five years post-publication
  Additional Notes:
  Data will be made available as soon as the primary results are published in a peer-reviewed journal.
  Access may be extended beyond five years based on research demand and institutional policies.
  Researchers requesting access must submit a formal data request and adhere to data-sharing agreements and ethical guidelines.
Access Criteria: Qualified researchers from academic, research, or healthcare institutions. Investigators conducting meta-analyses or related studies on PRF and alveolar preservation.
  Researchers with ethical approval and a valid research proposal.
  Available Data:
  De-identified CBCT images, clinical measurements (bone height, depth, HU values), demographic data (age, sex, health status), and outcome measures.
  Study protocol, data collection methods, and statistical analysis plan.
  Access Process:
  Submit a formal request detailing research objectives and ethics approval. Sign a data-sharing agreement to ensure ethical use and compliance. Secure data transfer via an encrypted institutional repository. This policy promotes research transparency, collaboration, and ethical data use while protecting participant privacy.

REFERENCES:
- [Background] Simon BI, Von Hagen S, Deasy MJ, Faldu M, Resnansky D. Changes in alveolar bone height and width following ridge augmentation using bone graft and membranes. J Periodontol. 2000 Nov;71(11):1774-91. doi: 10.1902/jop.2000.71.11.1774. PMID 11128929
- [Background] Anwandter A, Bohmann S, Nally M, Castro AB, Quirynen M, Pinto N. Dimensional changes of the post extraction alveolar ridge, preserved with Leukocyte- and Platelet Rich Fibrin: A clinical pilot study. J Dent. 2016 Sep;52:23-9. doi: 10.1016/j.jdent.2016.06.005. Epub 2016 Jun 20. PMID 27338946
- [Background] Alzahrani AA, Murriky A, Shafik S. Influence of platelet rich fibrin on post-extraction socket healing: A clinical and radiographic study. Saudi Dent J. 2017 Oct;29(4):149-155. doi: 10.1016/j.sdentj.2017.07.003. Epub 2017 Aug 2. PMID 29033524
- [Background] Hauser F, Gaydarov N, Badoud I, Vazquez L, Bernard JP, Ammann P. Clinical and histological evaluation of postextraction platelet-rich fibrin socket filling: a prospective randomized controlled study. Implant Dent. 2013 Jun;22(3):295-303. doi: 10.1097/ID.0b013e3182906eb3. PMID 23644909
- See also: The link contains forms used in the clinical trial on Platelet-Rich Fibrin (PRF) for alveolar preservation, including informed consent templates, clinical evaluation forms, radiographic analysis templates, and randomization records. Due to patient priva — https://ucacueedu-my.sharepoint.com/:f:/g/personal/rocio_molina_ucacue_edu_ec/EmUsBYq74wZGl8hxBeQ_cgYBc7hO98P4eFXFhnbsqcvzDw?e=WTIKei